CLINICAL TRIAL: NCT06420414
Title: Comparing Physiological and Psychological Effects of Virtual Reality Vs. Traditional HIIT In Healthy Individuals: Results From A Preliminary Pilot Randomised Controlled Trial
Brief Title: Physiological and Psychological Effects of Virtual Reality vs Traditional Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Jonathan Robinson, Ph.D, Senior Lecturer in Research Methods, Teesside University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10853
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Healthy; Physical Activity; Virtual Reality; Exergame; Inactivity, Physical
Keywords: Exergaming; Virtual Reality; Meta Oculus Quest; Heart rate; Rate of perceived exertion; Technology acceptance; Bayesian Inferences; Pilot; RCT; Healthy
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: This parallel-design pilot randomised controlled trial (RCT) had two arms, each representing a different intervention: one group used a virtual reality (VR) exergaming system ("FitXR" on the Facebook Oculus Quest 2) and the other performed traditional High-Intensity Interval Training (HIIT), mirroring the same movements and durations as in the VR game. Participants were allocated to the two arms via block randomisation, stratified by gender. Both groups underwent a 15-minute HIIT session with 10-second intervals, aimed at comparing physiological and psychological effects between VR and non-VR interventions.
Masking Description: The researcher who completed the data analysis (JR) was blinded to the participants and specifics of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (VR) HIIT (Experimental): Participants in this arm underwent a single session of High-Intensity Interval Training (HIIT) via the Facebook Oculus Quest 2 virtual reality headset and "FitXR" fitness game. This immersive VR environment engaged participants in a 15-minute HIIT session, involving squats, lunges, and punches to virtual targets. The intensity was comparable to traditional HIIT, with a 10-second rest between intervals.
  Interventions: Other: Virtual Reality
- Traditional HIIT (Active Comparator): Participants in this arm underwent a single session of traditional High-Intensity Interval Training (HIIT), mirroring the movements and duration of the "FitXR" VR game. Exercises like squats, lunges, and punching targets were replicated, ensuring the same 15-minute workout duration and 10-second rest intervals, as in the VR arm.
  Interventions: Other: Traditional HIIT

INTERVENTIONS:
Other: Virtual Reality — Participants engaged in a 15-minute HIIT session using the Facebook Oculus Quest 2 VR headset with the "FitXR" fitness game. The advanced level workout (High Speed) was chosen, where participants performed functional movements like squats, lunges, and trunk rotations while punching virtual targets. The VR environment provided a 10-second rest period between intervals and featured a virtual trainer's guidance.
  Other Names: Facebook Oculus Quest 2
  Arms: Virtual Reality (VR) HIIT
Other: Traditional HIIT — Participants followed a non-VR 15-minute HIIT programme designed to replicate the exercises and patterns seen in the "FitXR" game. The traditional exercises included squats, lunges, and punches, matching the VR programme's intensity and interval structure. Participants watched a pre-recorded video on a laptop, which guided them through the workout. The 10-second rest periods were also maintained for consistency.
  Arms: Traditional HIIT

SUMMARY:
This study aimed to explore the feasibility and effectiveness of immersive Virtual Reality (VR) as an alternative to traditional High-Intensity Interval Training (HIIT) by comparing physiological and psychological outcomes in physically active university students. The pilot randomised controlled trial utilised a parallel design involving two groups: one group performed HIIT using the Facebook Oculus Quest 2 VR headset with the "FitXR" fitness game, while the other undertook traditional HIIT training that mirrored the movements and actions of the VR game.

The study's findings suggest that fully immersive VR provides a unique and potentially more enjoyable alternative to traditional HIIT, particularly because it may enhance motivation while still achieving health benefits. This pilot research study highlights VR's potential to reach high-flow states in exercise, where individuals become deeply absorbed and derive satisfaction from the activity. It also lays the groundwork for future studies involving larger sample sizes and clinical populations to further investigate the psychological and physiological impacts of VR-based exercise.

In summary, this pilot randomised controlled trial found that immersive VR could be a feasible and effective alternative to traditional HIIT training, offering similar physiological benefits while enhancing exercise motivation and enjoyment. Further research is necessary to validate these preliminary results and extend them to diverse populations.

DETAILED DESCRIPTION:
Study Objectives and Design This study was designed as a pilot randomised controlled trial (RCT) to investigate the feasibility, efficacy, and effects of immersive VR compared to traditional HIIT on physiological and psychological outcomes in physically active university students. The parallel-design trial was conducted in accordance with the CONSORT guidelines and approved by the Teesside University Health Research Ethics Sub-Committee. The VR intervention used the Facebook Oculus Quest 2 VR headset with the fitness game "FitXR," while the non-VR group completed traditional HIIT that replicated the same movements as in the VR game.

Participants and Recruitment A purposive sampling method was used to recruit ten healthy physiotherapy students from Teesside University. Participants had to lead an active lifestyle, defined as performing either 150 minutes of moderate exercise weekly or 75 minutes of vigorous-intensity aerobic exercise, and have no prior experience with VR-based exercise. Those with medical conditions preventing them from exercising or those unable to give informed consent were excluded. Participants were recruited via email through a gatekeeper, indicating their willingness to participate by contacting the research physiotherapist directly. The allocation to either the VR or non-VR group was stratified by gender and block-randomised in blocks of five using a computer-generated software (Research Randomizer).

Interventions

Exergaming via VR:

Participants in the VR group used the Facebook Oculus Quest 2 and "FitXR," a fitness game in high-speed HIIT class mode. The 15-minute session included functional movements such as squats, lunges, and trunk rotations while trying to hit virtual targets by punching. The training session had a 10-second rest between each interval, and participants followed instructions from a virtual trainer.

Traditional HIIT:

The non-VR group followed a traditional HIIT session that mirrored the movements from the "FitXR" game. Participants replicated movements such as squats with punches, as pre-recorded and displayed on a laptop. The session matched the VR group's overall duration and intervals.

Safety and Blinding To ensure safety while using the VR headset, participants were restricted to a 3m by 3m safety boundary. Stepping out of the boundary automatically paused the game, activating external cameras to provide real-world visibility. Blinding was not feasible due to the nature of the intervention, but the researcher responsible for the data analysis was unaware of the group allocations to reduce bias.

Outcome Measures

Physiological Outcomes:

Heart Rate: Measured using a Polar RS400 monitor. Exercise intensity was calculated as a percentage of the maximum heart rate (%HRmax) and heart rate reserve (%HRR). The intensity was categorised according to American Heart Association standards.

Rating of Perceived Exertion (RPE): Measured using Borg's CR-10 scale every five minutes. Scores ranged from 0 (rest) to 10 (maximum effort).

Psychological Outcomes:

Flow State Scale (FSS): Assessed engagement and motivation using a 36-item questionnaire with nine subscales. Participants rated items on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). The subscales measured challenge-skill balance, action-awareness merging, clear goals, unambiguous feedback, and other factors.

Statistical Analysis A frequentist approach was employed with SPSS software (version 26). Independent-samples t-tests were used with a significance level of 0.05, and effect sizes were expressed using Cohen's d (small = 0.2, moderate = 0.5, large = 0.8). Bayesian data analysis was conducted with JASP software to assess the robustness of findings. Bayes factors were calculated to compare evidence for alternative versus null hypotheses. Robustness checks were performed to ensure results remained consistent across different prior distributions.

Sample Size and Feasibility Given that this was a pilot study, the emphasis was placed on assessing feasibility rather than ensuring the study was fully powered. As such, recruitment spanned a period of time with the objective of enrolling as many patients as possible, without specifying a target participant number to achieve optimal study power. An aim of this study was, therefore, to explore feasibility and preliminary outcomes, which will inform future, larger-scale research

Conclusion This pilot study provides preliminary evidence that immersive VR training can offer a feasible alternative to traditional HIIT, achieving comparable physiological benefits with potentially greater intrinsic motivation and engagement. Future studies with larger sample sizes are needed to validate these findings and assess VR's impacts on diverse clinical populations.

ELIGIBILITY:
Inclusion Criteria:

1. Teesside University physiotherapy student.
2. Participants willing and able to give informed consent.
3. Have an active lifestyle (performing either 150 minutes of moderate exercise weekly or 75 minutes of vigorous intensity aerobic exercise).
4. No prior experience with exercise using the VR headset.

Exclusion Criteria:

1. Have a known medical condition that would prevent them from exercising.
2. Are not able to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Heart Rate (HR) | During each 15-minute HIIT session for both VR and traditional groups.
  Average percentage of maximum heart rate (%HRmax) and heart rate reserve (%HRR), measured using the Polar HR monitor RS400. The intensity levels were classified according to American Heart Association guidelines: ≥50% HRmax or ≥45% HRR as moderate intensity and ≥70% HRmax or ≥60% HRR as vigorous intensity.
Perceived Exertion (RPE) | Every 5 minutes throughout the 15-minute HIIT session for both groups.
  Average score on the CR-10 BORG's scale, where 0 represents "rest" and 10 represents "maximal" effort. Perceived exertion scores were obtained every 5 minutes, and an average score was calculated. Higher scores are an indication of greater exertion.
Flow Experience | Immediately after each 15-minute HIIT session.
  The Flow State Scale (FSS) questionnaire measured the extent to which participants experienced flow states during their respective HIIT sessions. There is a total of 36 items with 9 subscales measuring challenge-skill balance, action awareness merging, clear goals, unambiguous feedback, concentration on the task at hand, paradox (or sense) of control, loss of self-consciousness, time transformation, and autotelic experience. Each question is measured using a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate a better outcome, reflecting a higher degree of flow experience.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Robinson, PhD, Principal Investigator — Teesside University
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No